CLINICAL TRIAL: NCT02952040
Title: Pharmacokinetic Study of ASP1517 - Evaluation of the Effect of Lanthanum Carbonate Hydrate on the Pharmacokinetics of ASP1517 in Non-elderly Healthy Adult Male Subjects -
Brief Title: A Drug Interaction Study to Evaluate the Pharmacokinetics of ASP1517 and Lanthanum Carbonate Hydrate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1517-CL-0205
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Healthy Subjects
Keywords: ASP1517; Pharmacokinetics; Drug-drug interaction
MeSH Terms: interventions — lanthanum carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP1517 alone period preceding group (Experimental): Subjects will receive a single oral dose of ASP1517 alone in period 1, then subjects will receive a single oral dose of ASP1517 with lanthanum carbonate hydrate in period 2.
  Interventions: Drug: ASP1517; Drug: Lanthanum carbonate hydrate
- ASP1517+lanthanum period preceding group (Experimental): Subjects will receive a single oral dose of ASP1517 with lanthanum carbonate hydrate in period 1, then subjects will receive a single oral dose of ASP1517 alone in period 2.
  Interventions: Drug: ASP1517; Drug: Lanthanum carbonate hydrate

INTERVENTIONS:
Drug: ASP1517 — Oral dose
Drug: Lanthanum carbonate hydrate — Oral dose
  Other Names: Fosrenol

SUMMARY:
The objective of this study is to evaluate the effect of lanthanum carbonate hydrate on the pharmacokinetics (PK) of ASP1517 in non-elderly healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body weight (at screening): ≥50.0 kg and <80.0 kg
* Body-mass index (at screening): ≥17.6 and <26.4 kg/m2 [Body-mass index = Body weight (kg)/(Height (m))2]
* Subject must agree to use contraception consisting of two established forms specified below starting at the time of informed consent and continuing throughout the treatment period and for 84 days after the last administration of ASP1517.
* Subject must agree not to donate sperm starting at the time of informed consent and continuing throughout 84 days after the last administration of ASP1517.

Exclusion Criteria:

* Received or is scheduled to receive any investigational drugs in other clinical trials or post-marketing studies within 120 days before screening or during the period from screening to the hospital admission day of the Period 1.
* Received or is scheduled to receive medications (including over-the-counter drugs) or supplements within 7 days before the hospital admission day of the Period 1.
* Deviates from any of the normal range of blood pressure, pulse rate, body temperature and standard 12-lead electrocardiogram at screening or the hospital admission day of the Period 1.
* Meets any of the following criteria for laboratory tests at screening or the hospital admission day of the Period 1. Normal ranges of each test specified at the study site or the test/assay organization will be used as the normal ranges in this study.
* Concurrent or previous drug allergies.
* Development of (an) upper gastrointestinal symptom(s) within 7 days before the hospital admission day of the Period 1.
* Concurrent or previous hepatic disease, heart disease, respiratory disease, peritoneum inflammation.
* A history of abdominal surgery, digestive tract excision.
* Concurrent or previous renal disease, endocrine disease, cerebrovascular disorder, malignant tumor, retinal neovascular lesions.
* Previous use of hypoxia inducible factor-prolyl hydroxylase inhibitors (HIF-PHI) such as ASP1517 (FG-4592), YM311 (FG-2216), erythropoietin products or lanthanum carbonate hydrate.
* Excessive alcohol or smoking habit.

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) parameter of ASP1517 in plasma: AUCINF | Up to 72hr after each dosing
  AUCinf: Area under the concentration-time curve from the time of dosing extrapolated to time infinity
PK parameter of ASP1517 in plasma: AUC24h | Up to 72hr after each dosing
  AUC24h: Area under the concentration-time curve from the time of dosing to 24h
PK parameter of ASP1517 in plasma: Cmax | Up to 72hr after each dosing
  Cmax: Maximum concentration

SECONDARY OUTCOMES:
PK parameter of ASP1517 in plasma: AUClast | Up to 72hr after each dosing
  AUC last: Area under the concentration-time curve from the time of dosing to the last measurable concentration
PK parameter of ASP1517 in plasma: CL/F | Up to 72hr after each dosing
  CL/F: Apparent total systemic clearance
PK parameter of ASP1517 in plasma: t1/2 | Up to 72hr after each dosing
  t1/2: Terminal elimination half-life
PK parameter of ASP1517 in plasma: Lambda z | Up to 72hr after each dosing
  Lambda z: Terminal elimination rate constant
PK parameter of ASP1517 in plasma: MRTinf | Up to 72hr after each dosing
  MRTinf: Mean residence time from the time of dosing extrapolated to time infinity
PK parameter of ASP1517 in plasma: tmax | Up to 72hr after each dosing
  tmax : Time of Cmax
PK parameter of ASP1517 in plasma: tlag | Up to 72hr after each dosing
  tlag: Time point prior to the time point corresponding to the first measurable (non-zero) concentration
PK parameter of ASP1517 in plasma: Vz/F | Up to 72hr after each dosing
  Vz/F: Apparent volume of distribution during the terminal elimination phase after single extra-vascular dosing
Safety assessed by incidence of adverse events | Up to 7 days after drug dosing of period 2
Safety assessed by supine blood pressure | Up to 7 days after drug dosing of period 2
Safety assessed by supine pulse rate | Up to 7 days after drug dosing of period 2
Safety assessed by axillary body temperature | Up to 7 days after drug dosing of period 2
Safety assessed by Laboratory tests: Hematology | Up to 7 days after drug dosing of period 2
Safety assessed by Laboratory tests: Blood biochemistry | Up to 7 days after drug dosing of period 2
Safety assessed by Laboratory tests: Urinalysis | Up to 7 days after drug dosing of period 2
Safety assessed by 12-lead electrocardiogram | Up to 7 days after drug dosing of period 2

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Site JP00001, Tokyo, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided